CLINICAL TRIAL: NCT03609424
Title: A Phase Ib/II Study of PDR001 Plus Imatinib for Metastatic or Unresectable GIST With Prior Failure of Imatinib, Sunitinib and Regorafenib
Brief Title: PDR001 Plus Imatinib for Metastatic or Unresectable GIST
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC1802
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — spartalizumab; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDR001 plus Imatinib (Experimental)
  Interventions: Drug: PDR001, Imatinib

INTERVENTIONS:
Drug: PDR001, Imatinib — -Phase Ib part
  : The standard 3+3 dose escalation scheme will be applied. DLTs will be evaluated during the first cycle (4 weeks).
  PDR001 400mg, every 4 weeks, IV
  Imatinib dose level -1 : 200mg, PO, QD Imatinib dose level 1 : 300mg, PO, QD Imatinib dose level 2 : 400mg, PO, QD
  -Phase II part
  * Recommended dose defined in phase Ib part will be tested

SUMMARY:
Assuming that PDR001, an anti-PD-1 antibody, with imatinib might be effective in advanced GIST after failure of standard TKI therapies including imatinib, sunitinib, and regorafenib. In this phase I/II study of PDR001 plus imatinib, it is aimed to evaluate the safety and efficacy of this regimen as 4th line of treatment in advanced GIST.

DETAILED DESCRIPTION:
Immunotherapy may be the novel strategy to enhance the outcomes of TKI-refractory GIST. Although current understanding of the immune response in GIST remains limited compared to other cancer types, several data suggest that the immunotherapy may be the way to overcome the mutation-related primary and secondary TKI resistance, and the exploration is needed.

The PD-1-PD-L1 pathway is the one of key targets for immune checkpoint inhibitor, and anti-PD-1 antibodies including pembrolizumab, nivolumab has already shown a remarkable efficacy in several cancer types including melanoma, lung cancer, and gastric cancer with approval by FDA in melanoma and lung cancer. PDR001 is a novel anti-PD-1 inhibitor under investigation for the treatment of multiple tumor types, and the available safety data from on-going clinical trials indicate that PDR001 monotherapy is generally well tolerated and the safety profile appears to be similar across different tumor types.

Recent phase II study reported that pembrolizumab, an anti-PD-1 inhibitor, demonstrated only modest anti-tumor efficacy in advanced GISTs. However, the sample size was small with only 10 GIST tumors in the study, and high proportion of GIST tumors were prominently infiltrated by IDO positive M2 macrophage, which plays important role in immune suppression. Thus, further strategies are warranted to assess the combination of immune checkpoint inhibitor with an agent which can inhibit the IDO pathway in advanced GIST.

PD-L1 expression has been regarded as a promising biomarker to predict the efficacy of anti-PD-1 or PD-L1 monoclonal antibodies, although negative PD-L1 expression do not preclude the efficacy of anti-PD-1 or PD-L1 antibodies. Although the data in regards to the PD-L1 expression in metastatic GISTs are limited, a recent study showed that the PD-L1 expression is observed in the subset of localized GIST tissue samples and its expression is correlated with prognosis. Further translational research of immune milieu using GIST tissues are necessary to establish the role of immunotherapy in metastatic GISTs, and concurrent prospective studies using immune check point inhibitors may enhance the speed of this work.

The relevance of continuous KIT inhibition in tyrosine kinase inhibitor (TKI) refractory GISTs was proven in previous phase III RIGHT study which compared imatinib rechallenge and placebo after failure of at least first line imatinib and second line sunitinib. In this study, the inhibition of KIT by imatinib was significantly associated with prolonged PFS (median PFS of 1.8 months) compared to placebo (median 0.9 month; HR 0.46, 95% CI 0.27-0.78; p=0.005). Disease control rate at 12 weeks was also improved with imatinib rechallenge than placebo (32% vs 5%, p=0.003).

Immune cells such as T cells (Treg), natural killer (NK) cells, and macrophages are present in GIST tissue samples, and their presence or activation were related with prognosis or response to imatinib. Imatinib indirectly have an impact on NK cells and CD8+ T cells, and concurrent use of CTLA-4 blockade with imatinib augments the efficacy of imatinib in mouse GIST by increasing IFN-r producing CD8+ T cells. Moreover, previous study showed that imatinib potentiates antitumor T-cell responses in GISTs through the inhibition of IDO. This may suggest that concurrent use of imatinib and immune checkpoint inhibitors may enhance the efficacy of immune checkpoint inhibitors.

Based on this background, we assume that PDR001, an anti-PD-1 antibody, with imatinib might be effective in advanced GIST after failure of standard TKI therapies including imatinib, sunitinib, and regorafenib. In this phase I/II study of PDR001 plus imatinib, It is aimed to evaluate the safety and efficacy of this regimen as 4th line of treatment in advanced GIST.

ELIGIBILITY:
1. Age 18 years or older, at the time of acquisition of informed consent
2. Histologically confirmed metastatic or unresectable GIST with CD117(+), DOG-1(+), or mutation in KIT or PDGFRαgene
3. Disease control (response or stabilization for at least 6 months) with first-line imatinib and failure (progression) to imatinib, sunitinib, and regorafenib. Disease progression is defined as (1) size increase ≥ 20% by RECIST version 1.1, (2) appearance of a definite new lesion (excluding small cystic new lesions in the liver within 6 months of starting TKIs), (3) new solid nodule ≥ at least 2 cm in size within a cystic mass, or (4) increase of the size ( ≥ 20%) of previously existing solid nodule ≥ at least 2 cm in size within a cystic mass.
4. ECOG performance status of 0-2
5. Resolution of all toxic effects of prior treatments to grade 0 or 1 by NCI-CTCAE version 4.0
6. At least one measurable lesion by RECIST version 1.1.
7. Adequate bone marrow, hepatic, renal, and other organ functions

   * Neutrophil ≥ 1,500/mm3
   * Platelet ≥ 75,000/mm3
   * Hemoglobin ≥ 8.0 g/dL
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * AST/ALT ≤ 3 x ULN without liver metastases or AST/ALT ≤ 5 x ULN with liver metastases
   * Creatinine≤ 1.5 x ULN
8. Women with reproductive potential must have a negative serum or urine pregnancy test
9. Washout period of previous TKIs or chemotherapy for more than 4 times the half-life (Seven days of washout period is enough for imatinib, sunitinib, and regorafenib).
10. No prior use of PDR001 or other immune check point inhibitors
11. Provision of a signed written informed consent

Exclusion criteria

1. Patients who are intolerant to imatinib
2. Women of child-bearing potential who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control.
3. Impaired cardiac function or clinically significant cardiac disease, including any of the following:

   Clinically significant and/or uncontrolled heart disease such as congestive heart failure (CHF) requiring treatment (NYHA grade ≥ 2), uncontrolled hypertension or clinically significant arrhythmia
   * Congenital long QT syndrome
   * QTc> 470 msec on screening ECG
   * Unstable angina pectoris ≤ 3 months prior to starting study drug
   * Acute Myocardial Infarction ≤ 3 months prior to starting study drug
4. Uncontrolled infection
5. History of severe hypersensitivity reactions to other monoclonal antibodies
6. Active autoimmune disease or a documented history of autoimmune disease, or any condition that requires systemic steroids, except vitiligo or resolved asthma/atopy that is treated with broncho-dilators (e.g., albuterol).
7. Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for this study
8. Major surgery ≤ 28 days prior to starting study drug or who have not recovered from side effects of such therapy
9. Known diagnosis of HIV infection (HIV testing is not mandatory)
10. History of another primary malignancy that is currently clinically significant or currently requires active intervention
11. Patients with brain metastases as assessed by radiologic imaging (e.g. CT, MRI) due to symptoms clinically suspected of brain metastases
12. Alcohol or substance abuse disorder
13. Active HBV and HCV infections requiring therapy: patients with undetectable HBV DNA level under the anti-viral agents are allowed to be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | up to 12 weeks
  Primary Outcome of phase Ib part
Recommended dose for expansion | up to 12 weeks
  Primary Outcome of phase Ib part
Disease control rate | up to 12 weeks
  Disease control rate (DCR: objective response + stable disease) at 12 weeks Primary Outcome of phase 2 part(defined by RECIST v1.1)

SECONDARY OUTCOMES:
Progression-free survival | Up to 2 years
  Progression-free survival (PFS) per the RECIST v1.1 and iRECIST PFS is defined as the time from the date of first dosing of PDR001 plus Imatinib to the date of progression or death due to any cause
Overall survival | Up to 2 years
  OS is defined as the time from the date of the start of PDR001 plus Imatinibto the time of death due to any cause
Response rate | Up to 2 years
  Response rate per the RECIST v1.1 and iRECIST Responses are assessed every 8 weeks (at fixed calendar time) until disease progression or death.
Toxicity profile | Up to 2 years
  Toxicity profile by the NCI-CTCAE v4.03
Correlation of efficacy with potential biomarkers | Up to 2 years
  Correlation of efficacy (DCR, ORR, PFS, and OS) with potential biomarkers including CD3, CD8, PD-1, PD-L1, LAG3, TIM3, CD204 (M2 macrophage), CD169 (M1 macrophage) using multiplex IHC
Mutational analysis | Up to 2 years
  Mutational analysis of KIT exons 9, 11, 13, and 17, and PDGFRα exons 12, 14, and 18 with direct sequencing using DNA extracted from archival tissues, newly obtained tissues at baseline, and/or at 4 weeks after the start of the study medication (biopsies at baseline and 4 weeks after study treatment are optional).

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea